CLINICAL TRIAL: NCT04626674
Title: An Open-Label, Systemic Gene Delivery Study Using Commercial Process Material to Evaluate the Safety of and Expression From SRP-9001 in Subjects With Duchenne Muscular Dystrophy (ENDEAVOR)
Brief Title: A Gene Transfer Therapy Study to Evaluate the Safety of and Expression From Delandistrogene Moxeparvovec (SRP-9001) in Participants With Duchenne Muscular Dystrophy (DMD)
Acronym: ENDEAVOR
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sarepta Therapeutics, Inc. (Industry)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SRP-9001-103
Record Dates: First submitted 2020-11-06; First posted 2020-11-12 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Muscular Dystrophy, Duchenne
Keywords: Duchenne Muscular Dystrophy; Gene-Delivery; DMD; Ambulatory Non-ambulatory; Pediatric; Dystrophin
MeSH Terms: conditions — Muscular Dystrophy, Duchenne

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Delandistrogene Moxeparvovec (Experimental): Participants will receive a single intravenous (IV) infusion of delandistrogene moxeparvovec on Day 1.
  Interventions: Genetic: delandistrogene moxeparvovec

INTERVENTIONS:
Genetic: delandistrogene moxeparvovec — Single IV infusion of delandistrogene moxeparvovec
  Other Names: SRP-9001; delandistrogene moxeparvovec-rokl; ELEVIDYS

SUMMARY:
This is an open-label gene transfer therapy study evaluating the safety of and expression from delandistrogene moxeparvovec in participants with DMD. The maximum participant duration for this study is 156 weeks.

ELIGIBILITY:
Inclusion Criteria:

* For Cohorts 1-8: Has a definitive diagnosis of DMD based on documented clinical findings and prior genetic testing.
* Cohort 1: Is ambulatory, and ≥4 to <8 years of age at the time of Screening.
* Cohort 2: Is ambulatory, and ≥8 to <18 years of age at the time of Screening.
* Cohort 3: Non-ambulatory per protocol specified criteria at the time of Screening.
* Cohort 4: Is ambulatory and ≥3 to <4 years of age at the time of Screening.
* Cohort 5a: Is ambulatory and ≥4 to <9 years of age with time to rise from the floor ≤7 seconds at the screening visit.
* Cohort 5b: Non-ambulatory per protocol specified criteria at the time of Screening.
* Cohort 6: Is ambulatory, and ≥2 to <3 years of age at the time of Screening.
* Cohort 7: Non-ambulatory per protocol-specified criteria at the time of Screening.
* Cohort 8: Non-ambulatory per protocol-specified criteria at the time of Screening, has a performance upper limb (PUL) entry item score ≥3 at the Screening visit and has a total PUL score of ≥20 and ≤40 at the time of Screening.
* Ability to cooperate with motor assessment testing.
* Cohorts 1, 2, 3, 5, 7 and 8 only: Stable dose equivalent of oral glucocorticoids for at least 12 weeks before screening and the dose is expected to remain constant (except for modifications to accommodate changes in weight) throughout the first year of the study.
* Cohorts 4 and 6: Do not yet require use of chronic steroids for treatment of their DMD, in the opinion of the Investigator, and are not receiving steroids at the time of Screening.
* rAAVrh74 antibody titers are not elevated as per protocol-specified requirements.
* Genetic mutation inclusion criteria vary by cohort.

Exclusion Criteria:

* Has a concomitant illness, autoimmune disease, chronic drug treatment, and/or cognitive delay/impairment that in the opinion of the Investigator creates unnecessary risks for gene transfer.
* Exposure to gene therapy, investigational medication, or any treatment designed to increase dystrophin expression within protocol-specified time limits.
* Abnormality in protocol-specified diagnostic evaluations or laboratory tests.
* Cohort 8: Any confounding factors that would prevent the use of oral sirolimus including a known hypersensitivity to sirolimus or any of its excipients.

Other inclusion/exclusion criteria apply.

Min Age: 2 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 83 (Estimated)
Dates: Start 2020-11-23 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-02-29 (Estimated)

PRIMARY OUTCOMES:
Part 1 (Cohorts 1 to 5): Change from Baseline in Quantity of Delandistrogene Moxeparvovec Dystrophin Expression at Week 12, as Measured by Western Blot | Baseline, Week 12
Part 1 (Cohorts 6 to 8): Quantity of Delandistrogene Moxeparvovec Dystrophin Expression at Week 12 as Measured by Western Blot | Week 12
Cohort 8: Number of Participants with Acute Liver Injury (ALI) | Baseline up to Week 72

SECONDARY OUTCOMES:
Vector Shedding, Measured in Urine, Saliva, and Stool Samples Post-Infusion | Day 1 up to Week 104
Level of Antibody Titers to Recombinant Adeno-Associated Virus Serotype rh74 (rAAVrh74) | Day 2 up to Week 156
Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Adverse Events of Special Interest (AESIs) | Baseline up to Week 156
Cohort 8: Number of Participants With Infections, Edema, Wound-healing Complications, Hyperlipidemia, Angioedema, and Intestinal Lung Disease/ Non-infectious Pneumonitis | Baseline up to Week 72
Change from Baseline in Quantity of Delandistrogene Moxeparvovec Dystrophin Protein Expression at Week 12, as Measured by Immunofluorescence (IF) Fiber Intensity | Baseline, Week 12
Change from Baseline in Quantity of Delandistrogene Moxeparvovec Dystrophin Protein Expression at Week 12, as Measured by IF Percent Dystrophin Positive Fibers (PDPF) | Baseline, Week 12
Quantity of Delandistrogene Moxeparvovec Dystrophin Protein Expression at Week 12 as Measured by IF Fiber Intensity | Week 12
Quantity of Delandistrogene Moxeparvovec Dystrophin Protein Expression at Week 12 as Measured by IF PDPF | Week 12
Cohort 8: Number of Participants With Hepatic AEs, Hepatic Biomarkers, and Laboratory Assessments Indicative of Either Acute Hepatocellular Injury or Acute Liver Dysfunction | Baseline up to Week 72
Cohort 8: Number of Participants with Severe ALI | Baseline up to Week 72
Cohort 8: Duration of Steroids Administered | Baseline up to Week 72

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Sarepta Therapeutics, Inc.
Locations (5):
- United States (5):
  - Stanford University, Palo Alto, California
  - University of California, Davis, Sacramento, California
  - Washington University in St. Louis, St Louis, Missouri
  - Nationwide Children's Hospital, Columbus, Ohio
  - Children's Hospital of The King's Daughters, Norfolk, Virginia

REFERENCES:
- [Derived] Potter RA, Moeller IH, Khan S, Haegel H, Hollenstein A, Steiner G, Wandel C, Murphy AP, Asher DR, Palatinsky E, Griffin DA, Mason S, Iannaccone ST, Zaidman CM, Rodino-Klapac LR. Immunologic investigations into transgene directed immune-mediated myositis following delandistrogene moxeparvovec gene therapy. Sci Rep. 2025 Jan 2;15(1):4. doi: 10.1038/s41598-024-84077-w. PMID 39747998
- [Derived] Zaidman CM, Proud CM, McDonald CM, Lehman KJ, Goedeker NL, Mason S, Murphy AP, Guridi M, Wang S, Reid C, Darton E, Wandel C, Lewis S, Malhotra J, Griffin DA, Potter RA, Rodino-Klapac LR, Mendell JR. Delandistrogene Moxeparvovec Gene Therapy in Ambulatory Patients (Aged >/=4 to <8 Years) with Duchenne Muscular Dystrophy: 1-Year Interim Results from Study SRP-9001-103 (ENDEAVOR). Ann Neurol. 2023 Nov;94(5):955-968. doi: 10.1002/ana.26755. Epub 2023 Sep 7. PMID 37539981